CLINICAL TRIAL: NCT06631196
Title: The Effect of Jacobson's Progressive Muscle Relaxation Technique on Anxiety and Fatigue Among Children With Leukemia Undergoing Chemotherapy.
Brief Title: Jacobson's Progressive Muscle Relaxation Technique on Children With Leukemia Undergoing Chemotherapy.
Acronym: JPMRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU-20-4-294 (IRB00013620)
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Leukemia; Children; Fatigue Related to Cancer Treatment; Anxiety
Keywords: Jacobson's Progressive Muscle Relaxation Technique; Anxiety; Fatigue; Children; Leukemia; Chemotherapy; nursing care
MeSH Terms: conditions — Leukemia; Anxiety Disorders; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): children will be subjected to standardized nursing care.
- Interventional group (Jacobson's PMRT) (Experimental): children will be subjected to the implementation of Jacobson's progressive muscle relaxation technique for children with leukemia undergoing chemotherapy.
  Interventions: Procedure: Jacobson's PMRT

INTERVENTIONS:
Procedure: Jacobson's PMRT — each child in the intervention group will perform five sessions of Jacobson's PMRT. Each session lasted for 15-20 minutes under the supervision of the researcher.
  Arms: Interventional group (Jacobson's PMRT)

SUMMARY:
The goal of this clinical trial is to determine the effect of Jacobson's progressive muscle relaxation technique on anxiety and fatigue among children with leukemia undergoing chemotherapy. The main research hypotheses are;

* Children with leukemia who receive Jacobson's progressive muscle relaxation technique exhibit less anxiety than those who don't receive it.
* Children with leukemia who receive Jacobson's progressive muscle relaxation technique exhibit less fatigue than those who don't receive it.

Researchers will compare Jacobson's progressive muscle relaxation technique with standardized nursing care on a child's anxiety and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with leukemia and received chemotherapy sessions.
* Age ranged from 7 to 15 years.

Exclusion Criteria:

* other disorders such as neurological diseases, cerebrovascular accidents, or mental illness.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale: | before and after intervention.
  This tool was developed initially by (Smets et al., 1995) to assess fatigue for the subject. The scale comprised 18 items and 3 subscales which are; General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue.
  The format, instructions, Likert response scale, and scoring method are identical to the PedsQL 4.0 Generic Core Scales, with higher scores indicating a better health-related quality of life (lower fatigue symptoms). A five-point Likert scale was used to evaluate the responses in which (zero= never a problem; one = almost never a problem; two= sometimes a problem; three= often a problem; four= almost always a problem). Items are reverse-scored and linearly transformed to a 0-100 scale as follows:
  * 0 = 100-76
  * 1 = 75-51
  * 2 = 50-26
  * 3 = 25-1
  * 4= 0

SECONDARY OUTCOMES:
Spence Children's Anxiety Scale - Child (SCAS-Child) | before and after intervention.
  This tool was developed initially by Spence, S.H., (1997) to assess the severity of anxiety symptoms for the subject. The scale consists of six subscales: Separation Anxiety, Social Phobia, Obsessive Compulsive Problems, Panic/Agoraphobia, Generalized Anxiety/Overanxious Symptoms and Fears of Physical Injury.
  Scores consist of a total raw score (range from 0 to 114) and six sub-scale scores, with higher scores indicating greater severity of anxiety symptoms. Sub-scales are computed by summing the following items:
  * Separation anxiety (items 5, 8, 12, 15, 16, 44)
  * Social phobia (items 6, 7, 9, 10, 29, 35)
  * Obsessive-compulsive (items 14, 19, 27, 40, 41, 42)
  * Panic/agoraphobia (items 13, 21, 28, 30, 32, 34, 36, 37, 39)
  * Physical Injury (items 2, 18, 23, 25, 33)
  * Generalized anxiety (items 1, 3, 4, 20, 22, 24) Items that are not scored in either the total score or the sub-scale scores are 11, 17, 26, 31, 38, 43, 45, and 46. They are not scored because they did

OTHER OUTCOMES:
Socio Demographic and Medical Data of Children with leukemia Undergoing Chemotherapy Structured Interview Schedule | before intervention
  This tool will be developed by the researcher to assess the socio-demographic and medical data of children undergoing chemotherapy. It will include 2 parts:
  Part I: Socio-demographic data: It includes age, gender, educational level, and residence.
  Part II: Medical data of children: It includes onset of disease, type of leukemia, prescribed chemotherapy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sulistyawati, E., Allenidekania, A., & Gayatri, D. (2021). Effect of progressive muscle relaxation on sleep quality and side effects of chemotherapy in children with cancer: randomized clinical trial. Open Access Macedonian Journal of Medical Sciences, 9(T4), 300-308. https://doi.org/10.3889/oamjms.2021.5774
- [Result] Pouraboli B, Poodineh Z, Jahani Y. The Effect of Relaxation Techniques on Anxiety, Fatigue and Sleep Quality of Parents of Children with Leukemia under Chemotherapy in South East Iran. Asian Pac J Cancer Prev. 2019 Oct 1;20(10):2903-2908. doi: 10.31557/APJCP.2019.20.10.2903. PMID 31653133
- [Result] Mohammed Ahmed Mohammed, E., Ali Ibrahim Almanzlawi, H., & Attia Abdel Naby Raslan, H. (2020). Effect of Progressive Muscle Relaxation on Pain and Fatigue among Post Cardiac Surgery Patients. Egyptian Journal of Health Care, 11(2), 736-745. https://doi:10.21608/ejhc.2020.180367
- [Result] Haggag, W, E., Soliman, H. (1997). The Arabic version of multidimensional fatigue inventory: reliability, validity and findings in three groups. Egyptian Journal of Psychiatry, 20(1), 85-97.
- [Result] Giri A, Tanaya K. (2019). Effect of Jacobson's progressive muscle relaxation exercise on anxiety among children diagnosed with leukemia admitted in selected hospital of Cuttack. International Journal of Health Sciences & Research, 9(2),151-155.
- [Result] Baccouche, K., Walha, A., Medhaffar, M., Kammoun, W., Ayadi, H., Moalla, Y., … Ghribi, F. (2017). Evaluation of Anxiety in Children with Acute Leukemia: A Prospective Study of 20 Cases. European Psychiatry, 41(S1), s131-s131. doi:10.1016/j.eurpsy.2017.01.1947
- [Result] Ali, N.S.( 2021). The Arabic version of Spence Children's Anxiety Scale - Child (SCAS-Child). Available from: https://www.scaswebsite.com/wp-content/uploads/2021/07/scas-child-arabic.pdf